CLINICAL TRIAL: NCT04815785
Title: A Multicenter, Prospective, Single-Arm, Objective Performance Criteria Study to Evaluate the Safety and Efficacy of TaurusOne® Transcatheter Aortic Valve System in Patients With Severe Calcific Aortic Stenosis
Brief Title: Safety and Efficacy of TaurusOne® Transcatheter Aortic Valve System in Patients With Severe Calcific Aortic Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other); General Hospital of Shenyang Military Region (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP12000-2
Record Dates: First submitted 2021-03-06; First posted 2021-03-25 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single set of test (Experimental): The experimental apparatus consisted of artificial aortic valve, transporter and loading system
  Interventions: Device: TaurusOne® transcatheter aortic valve replacement system

INTERVENTIONS:
Device: TaurusOne® transcatheter aortic valve replacement system — The TaurusOne® Transcatheter Aortic Valve System consists of an aortic valve, an associated delivery catheter and a loading system. The aortic valve consists of a self-expanding nitinol frame, a sealing skirt and valve leaflets, which are made of bovine pericardium. The delivery system is mainly composed of conical head, opacity ring, inner tube, top ring, middle tube, outer tube, booster rod, stress diffusion catheter, handle, etc. The outflow end of the aortic valve is provided with three fixing holes evenly distributed on the circumference on the top ring of the delivery catheter, so as to facilitate the installation, delivery and release of the aortic valve. Before the operation, the aortic valve needs to be installed into the sheath of the delivery catheter as required.

SUMMARY:
To observe and evaluate the safety and efficacy of TaurusOne® transcatheter aortic valve system in patients with severe calcific aortic stenosis through a prospective, multicenter clinical trial using objective performance criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily participate and sign the informed consent and are able to comply with the entire trial process;
* Age ≥ 70 years;
* Patients with severe calcific aortic stenosis confirmed by echocardiography (Transaortic flow velocity ≥ 4.0 m/s, or aortic-valve gradient ≥ 40 mmHg (1 mmHg = 0.133 kPa), or aortic valve area < 0.8 cm2, or effective orifice area < 0.5 cm2/m2);
* Patients who have symptoms obviously caused by aortic stenosis, NYHA Class II or worse;
* Patients who are unsuitable for conventional surgery evaluated by the cardiac team (including at least two cardiovascular surgeons) [13] *;
* Life expectancy after implantation of prosthetic valve is more than one year evaluated by the cardiac team (including at least two cardiac surgeons);
* Aortic annulus diameter ≥ 18 mm and ≤ 29 mm (measured by cardiac CT);
* Ascending aorta diameter < 50 mm

  *: If the patient meets any of the following criteria judged by a multidisciplinary cardiac team composed of cardiologists and cardiovascular surgeons, radiologists, anesthesiologists, etc. (at least two cardiovascular surgeons), the patient will be identified as unsuitable for conventional surgery (at least STS ≥ 8 points):
* Estimated risk of surgery-related death or disability > 50% within 1 year;
* ≥3 major organ damage that could not be improved by surgery;
* Obstacles related to surgical procedures judged as serious

Exclusion Criteria:

* Patients with bacteremia or toxemia;
* Previous endocarditis or active endocarditis;
* Acute myocardial infarction (Q-wave MI, or non-Q-wave MI with elevated creatine kinase isoenzyme and troponin T) within 30 days;
* Any intracardiac mass, left ventricular or atrial thrombus, vegetation on echocardiography;
* Symptomatic atrial fibrillation that cannot be improved by drug therapy;
* Familial hypertrophic cardiomyopathy;
* Mitral or tricuspid valve insufficiency (grade II regurgitation or higher);
* Previous aortic valve graft (mechanical or bioprosthetic valve);
* Known allergies to contrast agents, aspirin, heparin, ticlopidine drugs, nitinol shape memory alloy, or bovine products;
* Known contraindications or allergies to anticoagulant regimens, or inability to use anticoagulants throughout the trial;
* Other serious diseases that may reduce life expectancy to less than 12 months (such as clinically recurrent or metastatic cancer, congestive heart failure, etc.);
* Current substance abuse problems (e.g., alcohol, cocaine, heroin, etc.);
* Scheduled to undergo surgery that may result in protocol noncompliance or confounding in data interpretation.
* Cerebrovascular accident (CVA) in the past 6 months;
* Patients with common carotid artery or internal carotid artery or vertebral artery stenosis (>70%);
* White blood cell count <3×109/L, platelet count <50×109/L;
* Hemoglobin < 90 g/L;
* Patients with severe coagulopathy;
* Severe left ventricular dysfunction, left ventricular ejection fraction < 20%;
* Abdominal or thoracic aortic aneurysm;
* Hepatic encephalopathy or acute active hepatitis;
* On dialysis or baseline creatinine level > 2.5 mg/dL (221 μ mol/L);
* Bleeding tendency or history of coagulation disease or refusal of blood transfusion;
* Patients with active peptic ulcer or active gastrointestinal (GI) bleeding;
* Patients with neurological diseases that seriously affect mobility and activities of daily living;
* Patients with mental illness or psychological disorders who are unable to communicate effectively;
* Patients who need emergency surgery for any reason;
* Patients who have participated in other drug or medical device clinical trials within 3 months prior to screening;
* Other conditions that make the patient ineligible to participate in this clinical trial in judgement of investigators

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 12 months | 12 months
  All-cause mortality

SECONDARY OUTCOMES:
Device success rate (Immediate after procedure) | Immediate after procedure
  * Successful delivery and release of vascular access and prosthetic aortic valve, and successful withdrawal of the delivery catheter
  * Accurate placement of prosthetic aortic valve at the anatomical site
  * Prosthetic aortic valve meets the desired requirements (mean valve gradient < 20 mm Hg or maximal flow velocity < 3 m/s; No severe prosthetic valve regurgitation or perivalvular leak)
Procedure success rate | 72 hours after procedure/prior to discharge
  A successful procedure is defined as successful implantation of the prosthetic aortic valve at the correct anatomical site 72 hours after the operation or before discharge without severe prosthetic valve regurgitation or perivalvular leak.
Cardiac function improvement | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  NYHA functional classification

OTHER OUTCOMES:
Product performance evaluation | Immediate after procedure
  Product Performance includes grip loading, emptying , delivery, release, retrace, development and retrieval performance of delivery catheter system. Every item measured by:1=good 2=average 3=poor.
Operative complication | Immediately after procedure
  The rate of operative complication
The incidence of major adverse cardiovascular and cerebrovascular events during the trial(MACCEs) | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Incidence of MACCEs (mortality, stroke, myocardial infarction, and so on surgery, arrhythmias, conduction blocks) during the trial
Incidence of major adverse valve-related events (MAVREs) during the trial | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  including prosthetic valve-related death, permanent cardiac pacemaker implantation, permanent cardiac defibrillator implantation, prosthetic valve embolism, prosthetic valve thrombosis, prosthetic valve dysfunction.
hemorrhage | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Rate of patients with hemorrhage during the trial.
acute kidney injury | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Rate of patients with acute kidney injury during the trial.
Vascular Complications | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Vascular Complications
Other TAVI related complications | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Rate of patients with Other TAVI related complications during the trial. Other TAVI related complications include conversion to surgery, accidental cardiopulmonary mechanical assistance, coronary occlusion, ventricular septal perforation, mitral valve damage or loss of function, pericardial tamponade, endocarditis, valvular thrombosis, valvular ectopic (displacement, embolization, erroneous release), etc.
Valvular function | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Valvular function include valve stenosis, valve regurgitation, valve function (such as opening area, pressure gradient), perivalvular leakage, etc.
  There is Echo standard in VARC II to apply for valvular function assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peiga Medical Technology (Suzhou) Co., Ltd, Suzhou, Jiangsu, China